CLINICAL TRIAL: NCT00068302
Title: A Phase I Trial Of Sirolimus In Relapsed/Refractory Leukemia And Non-Hodgkin's Lymphoma
Brief Title: Sirolimus in Treating Young Patients With Relapsed or Refractory Acute Leukemia or Non-Hodgkin's Lymphoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Recruiting/enrolling participants halted prematurely but potentially will resume
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: National Childhood Cancer Foundation (Unknown); The Leukemia and Lymphoma Society (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000321392; CHP-755; CHP-IRB-2002-12-3086
Record Dates: First submitted 2003-09-10; First posted 2003-09-11 (Estimated); Last update posted 2015-03-12 (Estimated); Status verified 2013-07

CONDITIONS: Leukemia; Lymphoma
Keywords: recurrent childhood lymphoblastic lymphoma; recurrent childhood small noncleaved cell lymphoma; recurrent childhood large cell lymphoma; recurrent childhood acute myeloid leukemia; recurrent childhood acute lymphoblastic leukemia
MeSH Terms: conditions — Leukemia; Lymphoma; Burkitt Lymphoma; Dendritic Cell Sarcoma, Interdigitating; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sirolimus (Experimental): This is a dose escalation study including 4-dose levels. Subjects will receive a one-time loading dose of sirolimus on day 0, time 0. Subsequent dosing at the assigned dose level will start 24 hours following the initial loading dose
  Interventions: Drug: sirolimus

INTERVENTIONS:
Drug: sirolimus — 3-6 subjects will be enrolled into each dose level
  Other Names: rapamycin; Rapamune

SUMMARY:
RATIONALE: Drugs used in chemotherapy such as sirolimus use different ways to stop cancer cells from dividing so they stop growing or die.

PURPOSE: This phase I trial is studying the side effects and best dose of sirolimus in treating young patients with relapsed or refractory acute leukemia or non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of sirolimus in pediatric patients with refractory or relapsed acute leukemia or non-Hodgkin's lymphoma.
* Determine the dose-limiting toxic effects of this drug in these patients.
* Determine the trough levels produced by this drug in these patients.
* Determine the anti-leukemia/lymphoma activity of this drug in these patients.

OUTLINE: This is an open-label, dose-escalation study.

Patients receive oral sirolimus once daily on days 1-21. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of sirolimus until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

Patients are followed for survival.

PROJECTED ACCRUAL: A total of 3-30 patients will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed diagnosis of 1 of the following:

  * Acute lymphoblastic leukemia (ALL) OR acute myeloid leukemia (AML)

    * At least 25% blasts in the bone marrow
    * Recurrent or refractory disease
  * Non-Hodgkin's lymphoma (NHL)

    * Second or greater relapse as determined by physical or radiological evidence
* Disease for which there is no known curative therapy

PATIENT CHARACTERISTICS:

Age

* 21 and under

Performance status

* Karnofsky 50-100% (patients over 10 years of age)
* Lansky 50-100% (patients 10 years of age and under)

Life expectancy

* At least 4 weeks

Hematopoietic

* Absolute neutrophil count at least 1,000/mm^3*
* Platelet count at least 75,000/mm^3 (transfusion independent)*
* Hemoglobin at least 8.0 g/dL (may receive red blood cells (RBC) transfusions)* NOTE: *Patients with ALL, AML, and NHL with tumor metastatic to bone marrow, with granulocytopenia, anemia, and/or thrombocytopenia are eligible, but will not be evaluable for hematological toxicity

Hepatic

* Bilirubin no greater than 1.5 times normal
* alanine aminotransferase (ALT) no greater than 5 times normal
* Albumin at least 2 g/dL

Renal

* Creatinine based on age, as follows:

  * No greater than 0.8 mg/dL (5 years of age and under)
  * No greater than 1.0 mg/dL (6 to 10 years of age)
  * No greater than 1.2 mg/dL (11 to 15 years of age)
  * No greater than 1.5 mg/dL (over 15 years of age) OR
* Creatinine clearance or radioisotope glomerular filtration rate at least 70 mL/min

Cardiovascular

* Shortening fraction at least 28% by echocardiogram OR
* Ejection fraction at least 50% by gated radionuclide

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Able to ingest oral medication
* No known allergy to sirolimus, tacrolimus, or other mammalian target of rapamycin (mTOR) inhibitors
* No uncontrolled active infection

  * Fungal disease must be stable for at least 2 weeks prior to study entry
  * Documented negative blood cultures prior to study entry for patients with bacteremia
* No active graft-versus-host disease

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Recovered from prior immunotherapy
* More than 1 week since prior hematopoietic growth factors except for epoetin alfa
* At least 7 days since prior biologic antineoplastic agents
* At least 3 months since prior bone marrow or stem cell transplantation

Chemotherapy

* Recovered from all prior chemotherapy
* More than 2 weeks since prior myelosuppressive chemotherapy (4 weeks for nitrosoureas)
* Prior hydroxyurea within the past 2 weeks is allowed provided peripheral blast count has been stable or rising for at least 3 days

Endocrine therapy

* Prior corticosteroids within the past 2 weeks are allowed provided peripheral blast count has been stable or rising for at least 3 days

Radiotherapy

* Recovered from prior radiotherapy
* At least 2 weeks since prior local palliative radiotherapy
* At least 4 weeks since prior craniospinal radiotherapy or radiation to the pelvis of 50% or more
* At least 4 weeks since prior substantial bone marrow radiotherapy
* No concurrent radiotherapy, except for emergent situations or persistent extramedullary disease with resolution of bone marrow disease

Surgery

* Not specified

Other

* No other concurrent investigational antineoplastic drugs
* No concurrent administration of any of the following:

  * Ketoconazole
  * Tacrolimus
  * Cyclosporine
  * Rifampin
  * Diltiazem

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2003-01; Primary Completion 2009-04 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Toxicity as assessed by Common Toxicity Criteria (CTC) toxicity criteria after the first course of treatment | within 21 days following administration of sirolimus
  Subjects will be assessed for toxicity on days 3, 7 and 21

SECONDARY OUTCOMES:
Response as assessed by radiologic scans after each course of treatment | day 21
  Response will be assessed on day 21 of cycle 1

CONTACTS AND LOCATIONS:
Overall Officials: Susan Rheingold, MD, Study Chair — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States